CLINICAL TRIAL: NCT02145117
Title: Neuroimaging Biomarkers of Mind-Body Treatment in Veterans With Post Traumatic Headache (PTH)
Brief Title: Brain Biomarkers w/Mind-Body Tx in Veterans With Post Traumatic Headache (PTH)
Acronym: MBSR-PTH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: VA Medical Center-West Los Angeles (U.S. Federal Agency); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Kirsten Tillisch, MD, MD, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-000864; R01AT007137 (NIH)
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Post Traumatic Headache
Keywords: MBSR; fMRI; PTH
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MBSR Training (Other): Mindfulness Based Stress Reduction (MBSR) Training
  Interventions: Behavioral: MBSR

INTERVENTIONS:
Behavioral: MBSR — Behavioral
  Other Names: Mindfullness Based Stress Reduction Training

SUMMARY:
This project aims to develop and test structural and functional brain imaging biomarkers for improvement in chronic pain from a mind/body intervention perspective in a critical veteran population, namely veterans with post traumatic headache (PTH) associated with mild traumatic brain injury (TBI). The project also aims to examine feasibility in a sample of veterans with PTH of performing resting state and structural neuroimaging protocols, and of obtaining active participation and completion of MBSR training. Lastly, exploratory analysis of brain imaging data will be performed to determine if hypothesized candidate biomarkers are associated with positive outcomes from MBSR and determine estimated effect sizes for future studies in PTH population.

DETAILED DESCRIPTION:
Returning veterans from Iraq and Afghanistan (OIF/OEF veterans) have a very high incidence of TBI (14-23%) with the largest number having mild TBI (i.e., no discernible structural brain damage) with 63.5% having persistent headache. Treatment of PTH in this population has been difficult and mind/body interventions including Mindfulness Based Stress Reduction (MBSR) may offer significant benefit. A biomarker that will support clinical endpoints ("surrogate endpoint") and help predict clinical benefit, could be used to more efficiently and completely assess mind/body treatment effects in clinical trials for PTH, compare various complementary and alternative medicine (CAM) treatments, and potentially target specific treatments to patients most likely to benefit. This project aims to investigate candidate biomarkers for MBSR response in veterans with PTH. Primarily, all subjects if they are interested and appropriate for the study, will undergo a screening at their regular clinic visit at the VAGLAS physical medicine and rehab department. If a subject responds to advertisement they will be screened using the same tools and enrollment criteria required for the veterans at VAGLAS. We expect we will need to enroll and screen no less than 33 subjects in order to complete 20 evaluable subjects for analysis. The study subjects will be evaluated for the severity of their PTH, the impact of PTH on their life, and the extent of the disease/pain condition. If eligible the nurse coordinator will contact them to schedule the pre-MBSR functional MRI visit. At the MRI we will evaluate patterns of activity (functional connectivity) in the brain at rest, and look at cortical thickness. Following the MRI visit all subjects will complete a 9-week modified MBSR training with a qualified instructor. Mid-study (after MBSR class 4) the subject will be asked to complete mid-study questionnaires at home on Survey Monkey or on paper if they choose. At the end of the MBSR training in which the subject will have to complete at least 3 visits, functional (f)MRI procedure will be repeated and compared against the first. Three months after completing the study there will be a follow-up visit to complete behavioral/symptom/quality of life questionnaires on line via SurveyMonkey. This is to see if the changes in the biomarkers will mediate changes in these behavioral measures 3-mo post Treatment (i.e. measure stability).

All in all, to complete the study subjects will have a screening visit, pre and post training MRI visit, up to 9 MBSR training visits, mid study questionnaires, a 4-hr retreat visit after week 6 and a final 3-mo f/u visit for questionnaires only.

ELIGIBILITY:
Inclusion Criteria:

* Males and female veterans at least 18 years of age
* Mild post traumatic headaches, diagnosed by a physician
* No prior training in MBSR or other mindfulness or meditation training will be allowed
* Able to read and speak English
* No participation in a clinical trial within the last 28 days

Exclusion Criteria:

* Current severe psychiatric diagnoses (e.g., schizophrenia, bipolar disorder, claustrophobia, history of panic attacks)
* Significant co-morbid condition(s) such as insulin-dependent diabetes, cancer, obesity (BMI>35), severe lung disease, neurological conditions (e.g., seizures), uncontrolled hypertension, or significant heart disease
* History of persistent headaches prior to TBI
* Unsafe for MRI (e.g., metal objects/shrapnel, metallic implants, brain or skull abnormalities, and claustrophobia)
* Use of centrally acting medications that will interfere with the neuroimaging testing (e.g. narcotic medications)
* Daily use of illicit drugs or marijuana
* Daily alcohol consumption of greater than 2 units

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-09; Primary Completion 2018-09-27 (Estimated); Study Completion 2018-09-27 (Estimated)

PRIMARY OUTCOMES:
Validate Optimal Biomarker candidates | After MBSR training (9 weeks)
  To validate optimal brain biomarker candidates by assessment of treatment responsiveness in post traumatic headache following a 9 week course in Mindfulness Based Stress Reduction (MBSR)

SECONDARY OUTCOMES:
Specificity, generality and moderation of biomarker response to MBSR treatment | Post MBSR training at 3 month follow up
  Specificity of biomarker response to MBSR measured by changes in selected biomarker candidates correlation with improvement in mindfulness at end of treatment and 3-month follow-up.
  Determine generality of optimal biomarkers via examination of factors such as sex, age, co-morbid pain, mood, and/or baseline severity, as moderators of biomarker performance.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Tillisch, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- VA West Los Angeles Medical Center, Los Angeles, California, United States